CLINICAL TRIAL: NCT04387565
Title: Analysis of Maternal Plasma/Urine/Hair Magnesium and Vanadium Levels in Preeclampsia (PrE)
Brief Title: Magnesium and Vanadium Levels in Preeclampsia
Acronym: V-Mg&PrE
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH7
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, urine, and hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preeclampsia: The diagnosis of LOPE, as will be defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), will be established based on the presence of proteinuria and a blood pressure level of ≥140/90 mmHg that occurs after 34 weeks of gestation in a previously normotensive woman. The diastolic and/or systolic blood pressure ≥ 160/110 mm Hg, it will be accepted as mild; and in case these values exceeded this level, it will be accepted as severe.
  Interventions: Other: magnesium and vanadium measurements and compare
- control pregnant group: These participants with normal healthy pregnancies at the third trimester (before birth)
  Interventions: Other: magnesium and vanadium measurements and compare
- control non-pregnant group: A volunteer group of healthy women who visited the gynaecology clinic for routine examinations and women who were admitted for pre-pregnancy tests were invited randomly to this research as a control group.
  Interventions: Other: magnesium and vanadium measurements and compare

INTERVENTIONS:
Other: magnesium and vanadium measurements and compare — Magnesium and vanadium will be measured using inductively coupled plasma-mass spectrometry (Thermo Scientific ICAPQc, USA).

SUMMARY:
Introduction: Vanadium important pollutants produced from anthropogenic activities, has been suggested to be embryotoxic and fetotoxic in a lot of studies. Magnesium sulfate therapy is used very common to prevent seizures in women with preeclampsia. However, the causes of preeclampsia are little known and heavy metals merit further investigation. The investigators will be tested whether late - onset preeclampsia (LOPE) was associated with exposure to these metals.

Methods: This study was designed to determine maternal plasma/urine/hair magnesium and vanadium concentrations in women with LOPE (n=70) compared to those of normotensive pregnant women (n=70) and to those of normotensive-healthy non-pregnant women (n=70). These metals concentrations will be measured using inductively coupled plasma-mass spectrometry were compared.

DETAILED DESCRIPTION:
This observational case-control study will be conducted at the Department of Obstetrics and Gynecology, Cengiz Gokcek Public Hospital, Gaziantep, Turkey, between May 2020 and February 2021. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (reference no: 2020/130). The study strictly will be adhered to the principles of the Declaration of Helsinki. All participants will be included in the study gave oral and written informed consent. Two-hundred ten women will be enrolled in the study in three groups.

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia
* healthy pregnancy
* healthy women

Exclusion Criteria:

1. pregnant women with any systemic condition (such as chronic hypertension, renal disease and diabetes mellitus)
2. using any kind of medication/supplement intake throughout pregnancy (such as heparin)
3. history of medication for PE treatment at the time of first admission
4. smoking
5. drug user
6. patients who had fetal congenital abnormalities or genetic syndromes
7. multiple-gestation pregnancies
8. pregnancies resulting from in vitro fertilization
9. intrauterine fetal death
10. having a family history of preeclampsia
11. Women who have menstrual irregularity
12. Women who have dyed their hair in the last 9 months
13. Gestational diabetes mellitus
14. Women receiving vanadium and/or magnesium treatment

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: The investigators consecutively will be recruited 70 late-onset preeclampsia patients as a study group, 70 participants with normal pregnancies as control pregnant group and 70 participants with healthy volunteer women as control non-pregnant group.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
magnesium and vanadium levels | 10 day
  The primary outcome in these analyses will be magnesium and vanadium levels in LOPE group and control groups.

SECONDARY OUTCOMES:
magnesium and vanadium levels in severy LOPE group | 1 day
  The secondary outcome will be compare the magnesium and vanadium levels in mild LOPE group and severy LOPE group.

OTHER OUTCOMES:
magnesium and vanadium levels in SGA group | 1 day
  Tertiary outcome will be compared the magnesium and vanadium levels in SGA group and non-SGA group.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ovayolu, MD, Principal Investigator — Cengiz Gökçek Kadın Doğum Ve Çocuk Hastalıkları Hastanesi
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ovayolu A, Ovayolu G, Karaman E, Yuce T, Ozek MA, Turksoy VA. Amniotic fluid levels of selected trace elements and heavy metals in pregnancies complicated with neural tube defects. Congenit Anom (Kyoto). 2020 Sep;60(5):136-141. doi: 10.1111/cga.12363. Epub 2019 Nov 27. PMID 31743503
- [Result] Scibior A. Vanadium (V) and magnesium (Mg) - In vivo interactions: A review. Chem Biol Interact. 2016 Oct 25;258:214-33. doi: 10.1016/j.cbi.2016.09.007. Epub 2016 Sep 13. PMID 27620816
- [Result] Elongi Moyene JP, Scheers H, Tandu-Umba B, Haufroid V, Buassa-Bu-Tsumbu B, Verdonck F, Spitz B, Nemery B. Preeclampsia and toxic metals: a case-control study in Kinshasa, DR Congo. Environ Health. 2016 Apr 5;15:48. doi: 10.1186/s12940-016-0132-1. PMID 27044488
- [Result] Euser AG, Cipolla MJ. Magnesium sulfate for the treatment of eclampsia: a brief review. Stroke. 2009 Apr;40(4):1169-75. doi: 10.1161/STROKEAHA.108.527788. Epub 2009 Feb 10. PMID 19211496
- [Result] Jiang M, Li Y, Zhang B, Zhou A, Zheng T, Qian Z, Du X, Zhou Y, Pan X, Hu J, Wu C, Peng Y, Liu W, Zhang C, Xia W, Xu S. A nested case-control study of prenatal vanadium exposure and low birthweight. Hum Reprod. 2016 Sep;31(9):2135-41. doi: 10.1093/humrep/dew176. Epub 2016 Jul 4. PMID 27381766
- [Derived] Ovayolu A, Turksoy VA, Turan AI, Dogan I, Bostancieri N. Does magnesium, one of the treatments for preeclampsia, interact with vanadium? Naunyn Schmiedebergs Arch Pharmacol. 2025 Sep 29. doi: 10.1007/s00210-025-04609-7. Online ahead of print. PMID 41020941

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04387565/Prot_SAP_000.pdf